CLINICAL TRIAL: NCT06647433
Title: What is the Perceived Role of Risk in the Healthcare Received by People in Disorders of Consciousness (DOC)?
Brief Title: What is the Perceived Role of Risk in DOC Healthcare.
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Royal Hospital for Neuro-disability (Other)
Responsible Party: Sponsor
Other Study IDs: 24051
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Disorders of Consciousness
Keywords: Disorders of Consciousness; Decision making
MeSH Terms: conditions — Consciousness Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — case study will be observed participants, methods will include observation, interview and video reflexive ethnography

SUMMARY:
Critical ethnography exploring how decisions are made on behalf of people in disorder of consciousness (DOC).

Prospective longitudinal case study design including observation, field interview and video reflexive ethnography.

ELIGIBILITY:
Inclusion Criteria:

* People in a DOC:
* Working diagnosis of being in a DOC.
* Have an appropriate family member able to act as a consultee.
* Over 18 years of age.

Family members and healthcare workers:

* conversational English.
* able to give consent.
* over 18 years of age.
* Involved in decision making on behalf of a person in a DOC

Exclusion Criteria:

Person in a Disorder of Consciousness

* Not in a DOC, diagnosis uncertain, or appears to be emerging.
* Clinically unstable or approaching the end of their life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people in a doc
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Meaning based themes on what influences decision making in DOC | 2 years
  Thematic analysis (TA) will consolidate and develop themes across all data sources (i.e., interview and VRE transcripts, field notes). The planned TA approach will borrow theory from reflexive thematic analysis (Braun & Clarke, 2022) and a critical realist TA approach which supports causal explanation development (Fryer, 2022). Causal research questions will be developed and refined throughout data collection and explored through TA.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Hospital for Neurodisability, London, London
  - University of Nottingham, Nottingham